CLINICAL TRIAL: NCT03763708
Title: Spinal Cord Stimulation Research Study
Brief Title: SCS Research Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business temporarily suspended study January 2023 with intent to include additional cohorts in future. For business reasons, study terminated April 2024.
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT18036
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Results first posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Limb Pain; Trunk Pain
MeSH Terms: interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (9):
- Cohort 1: Low Energy - Continuous (Experimental): Subjects will be programmed to a specific frequency with a long pulse width at various amplitudes
  Interventions: Device: Spinal Cord Stimulation
- Cohort 2: Interleaving (Experimental): Determine effects of delivering ping pulses combined with governed pulses while using separate sets of electrodes
  Interventions: Device: Spinal Cord Stimulation
- Cohort 3: Cycling Evolve (Experimental): Subjects will be programmed to high dose (HD) stimulation with various cycling parameters
  Interventions: Device: Spinal Cord Stimulation
- Cohort 4: Low Energy Cycling 1 (Experimental): Effects of decreased pulse widths with increased frequency - with and without cycling parameters
  Interventions: Device: Spinal Cord Stimulation
- Cohort 5: Low Energy Cycling 2 (Experimental): Effects of decreased pulse widths with increased frequency - with and without cycling parameters (different pulse widths and frequencies than Cohort 4)
  Interventions: Device: Spinal Cord Stimulation
- Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS) (Experimental): Effects of decreased frequency and therapy cycling parameters
  Interventions: Device: Spinal Cord Stimulation
- Cohort 7: Super Cycle (Experimental): Effects of longer cycle duration
  Interventions: Device: Spinal Cord Stimulation
- Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS) (Experimental): Effects of integrating Neuro Sense into DTM programming
  Interventions: Device: Spinal Cord Stimulation
- Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow (Experimental): Characteristics of vital signs in DPN participants
  Interventions: Device: Spinal Cord Stimulation

INTERVENTIONS:
Device: Spinal Cord Stimulation — Programming

SUMMARY:
To characterize the effects of stimulation parameters on pain relief and other cohort specific outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. 22 years of age or older
2. Implanted with a Medtronic rechargeable neurostimulation system, for a labeled indication, for at least 1 month and expected longevity of neurostimulator is at least 5 months
3. Willing and able to provide signed and dated informed consent
4. Capable of comprehending and consenting in English
5. Willing and able to comply with all study procedures, including diary completion, and visits
6. Able to differentiate between pain associated with the indication for SCS implant and other types of pain

Exclusion Criteria:

1. Implanted with neurostimulation system for an off-label indication
2. Currently enrolled or planning to enroll in an interventional clinical study that could potentially confound the study results
3. If female, pregnant or is of child-bearing potential and unwilling to use a medically acceptable form of birth control during the study
4. Has untreated major psychiatric comorbidity
5. Has a non-rechargeable neurostimulator where the battery longevity is not able to be estimated with the battery longevity calculator

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Center for Pain and Supportive Care, Phoenix, Arizona
  - Goodman Campbell Brain and Spine, Carmel, Indiana
  - Drez One, Somerset, Kentucky
  - Twin Cities Pain Clinic, Edina, Minnesota
  - Regional Brain and Spine, Cape Girardeau, Missouri
  - Carolinas Research Institute, Huntersville, North Carolina
  - Center for Interventional Pain and Spine, Lancaster, Pennsylvania
  - Pain Diagnostics and Interventional Care, Sewickley, Pennsylvania
  - Northwest Pain Care, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some subjects participated in more than one cohort during the lifecycle of the study.
Period: Cohort 1: Low Energy -Continuous
Arm/Group | Cohort 1: Low Energy - Continuous | Cohort 2: Interleaving | Cohort 3: Cycling Evolve | Cohort 4: Low Energy Cycling 1 | Cohort 5: Low Energy Cycling 2 | Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS) | Cohort 7: Super Cycle | Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS) | Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow
Started | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 2: Interleaving
Arm/Group | Cohort 1: Low Energy - Continuous | Cohort 2: Interleaving | Cohort 3: Cycling Evolve | Cohort 4: Low Energy Cycling 1 | Cohort 5: Low Energy Cycling 2 | Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS) | Cohort 7: Super Cycle | Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS) | Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow
Started | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 3: Cycling Evolve
Arm/Group | Cohort 1: Low Energy - Continuous | Cohort 2: Interleaving | Cohort 3: Cycling Evolve | Cohort 4: Low Energy Cycling 1 | Cohort 5: Low Energy Cycling 2 | Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS) | Cohort 7: Super Cycle | Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS) | Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow
Started | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 4: Low Energy Cycling 1
Arm/Group | Cohort 1: Low Energy - Continuous | Cohort 2: Interleaving | Cohort 3: Cycling Evolve | Cohort 4: Low Energy Cycling 1 | Cohort 5: Low Energy Cycling 2 | Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS) | Cohort 7: Super Cycle | Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS) | Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow
Started | 0 | 0 | 0 | 15 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 13 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Period: Cohort 5: Low Energy Cycling 2
Arm/Group | Cohort 1: Low Energy - Continuous | Cohort 2: Interleaving | Cohort 3: Cycling Evolve | Cohort 4: Low Energy Cycling 1 | Cohort 5: Low Energy Cycling 2 | Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS) | Cohort 7: Super Cycle | Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS) | Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow
Started | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 13 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Period: Cohort 6: DTM-LE SCS
Arm/Group | Cohort 1: Low Energy - Continuous | Cohort 2: Interleaving | Cohort 3: Cycling Evolve | Cohort 4: Low Energy Cycling 1 | Cohort 5: Low Energy Cycling 2 | Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS) | Cohort 7: Super Cycle | Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS) | Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow
Started | 0 | 0 | 0 | 0 | 0 | 22 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 20 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Period: Cohort 7: Super Cycle
Arm/Group | Cohort 1: Low Energy - Continuous | Cohort 2: Interleaving | Cohort 3: Cycling Evolve | Cohort 4: Low Energy Cycling 1 | Cohort 5: Low Energy Cycling 2 | Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS) | Cohort 7: Super Cycle | Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS) | Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow
Started | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Screen Failure | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Cohort 8: DTM for NS
Arm/Group | Cohort 1: Low Energy - Continuous | Cohort 2: Interleaving | Cohort 3: Cycling Evolve | Cohort 4: Low Energy Cycling 1 | Cohort 5: Low Energy Cycling 2 | Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS) | Cohort 7: Super Cycle | Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS) | Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 9: DPN Flow
Arm/Group | Cohort 1: Low Energy - Continuous | Cohort 2: Interleaving | Cohort 3: Cycling Evolve | Cohort 4: Low Energy Cycling 1 | Cohort 5: Low Energy Cycling 2 | Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS) | Cohort 7: Super Cycle | Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS) | Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Screen Failure | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Some participants were in more than one cohort; total enrollment is 100 participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Low Energy - Continuous | Cohort 2: Interleaving | Cohort 3: Cycling Evolve | Cohort 4: Low Energy Cycling 1 | Cohort 5: Low Energy Cycling 2 | Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS) | Cohort 7: Super Cycle | Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS) | Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow | Total
Number analyzed (Participants) | 15 | 10 | 4 | 15 | 15 | 22 | 17 | 4 | 11 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Some participants joined a new cohort once their current cohort was completed, and they met the new cohort guidelines. Therefore, there were participants who ended up in more than one of the 9 cohorts. There were a total of 100 unique participants in this study.
  years
    Cohort 1: Low Energy - Continuous: number analyzed (Participants) | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15
    Cohort 1: Low Energy - Continuous | 60.5 (7.9) |  |  |  |  |  |  |  |  | 60.5 (7.9)
    Cohort 2: Interleaving: number analyzed (Participants) | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10
    Cohort 2: Interleaving |  | 55.6 (9.5) |  |  |  |  |  |  |  | 55.6 (9.5)
    Cohort 3: Cycling Evolve: number analyzed (Participants) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 4
    Cohort 3: Cycling Evolve |  |  | 59.4 (9.0) |  |  |  |  |  |  | 59.4 (9.0)
    Cohort 4: Low Energy Cycling 1: number analyzed (Participants) | 0 | 0 | 0 | 15 | 0 | 0 | 0 | 0 | 0 | 15
    Cohort 4: Low Energy Cycling 1 |  |  |  | 55.0 (10.5) |  |  |  |  |  | 55.0 (10.5)
    Cohort 5: Low Energy Cycling 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 0 | 0 | 15
    Cohort 5: Low Energy Cycling 2 |  |  |  |  | 55.2 (12.3) |  |  |  |  | 55.2 (12.3)
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 22 | 0 | 0 | 0 | 22
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS) |  |  |  |  |  | 62.4 (11.4) |  |  |  | 62.4 (11.4)
    Cohort 7: Super Cycle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 0 | 17
    Cohort 7: Super Cycle |  |  |  |  |  |  | 64.9 (8.7) |  |  | 64.9 (8.7)
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 4
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS) |  |  |  |  |  |  |  | 66.25 (17.3) |  | 66.25 (17.3)
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow |  |  |  |  |  |  |  |  | 55.9 (16.37) | 55.9 (16.37)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Some participants joined a new cohort once their current cohort was completed, and they met the new cohort guidelines. Therefore, there were participants who ended up in more than one of the 9 cohorts. There were a total of 100 unique participants in this study.
  Participants
    Cohort 1: Low Energy - Continuous: number analyzed (Participants) | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15
    Cohort 1: Low Energy - Continuous: Female | 8 |  |  |  |  |  |  |  |  | 8
    Cohort 1: Low Energy - Continuous: Male | 7 |  |  |  |  |  |  |  |  | 7
    Cohort 2: Interleaving: number analyzed (Participants) | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10
    Cohort 2: Interleaving: Female |  | 6 |  |  |  |  |  |  |  | 6
    Cohort 2: Interleaving: Male |  | 4 |  |  |  |  |  |  |  | 4
    Cohort 3: Cycling Evolve: number analyzed (Participants) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 4
    Cohort 3: Cycling Evolve: Female |  |  | 2 |  |  |  |  |  |  | 2
    Cohort 3: Cycling Evolve: Male |  |  | 2 |  |  |  |  |  |  | 2
    Cohort 4: Low Energy Cycling 1: number analyzed (Participants) | 0 | 0 | 0 | 15 | 0 | 0 | 0 | 0 | 0 | 15
    Cohort 4: Low Energy Cycling 1: Female |  |  |  | 5 |  |  |  |  |  | 5
    Cohort 4: Low Energy Cycling 1: Male |  |  |  | 10 |  |  |  |  |  | 10
    Cohort 5: Low Energy Cycling 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 0 | 0 | 15
    Cohort 5: Low Energy Cycling 2: Female |  |  |  |  | 7 |  |  |  |  | 7
    Cohort 5: Low Energy Cycling 2: Male |  |  |  |  | 8 |  |  |  |  | 8
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 22 | 0 | 0 | 0 | 22
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Female |  |  |  |  |  | 13 |  |  |  | 13
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Male |  |  |  |  |  | 9 |  |  |  | 9
    Cohort 7: Super Cycle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 0 | 17
    Cohort 7: Super Cycle: Female |  |  |  |  |  |  | 10 |  |  | 10
    Cohort 7: Super Cycle: Male |  |  |  |  |  |  | 7 |  |  | 7
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 4
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): Female |  |  |  |  |  |  |  | 1 |  | 1
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): Male |  |  |  |  |  |  |  | 3 |  | 3
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: Female |  |  |  |  |  |  |  |  | 6 | 6
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: Male |  |  |  |  |  |  |  |  | 5 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Some participants joined a new cohort once their current cohort was completed, and they met the new cohort guidelines. Therefore, there were participants who ended up in more than one of the 9 cohorts. There were a total of 100 unique participants in this study.
  Participants
    Cohort 1: Low Energy - Continuous: number analyzed (Participants) | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15
    Cohort 1: Low Energy - Continuous: Hispanic or Latino | 0 |  |  |  |  |  |  |  |  | 0
    Cohort 1: Low Energy - Continuous: Not Hispanic or Latino | 15 |  |  |  |  |  |  |  |  | 15
    Cohort 1: Low Energy - Continuous: Unknown or Not Reported | 0 |  |  |  |  |  |  |  |  | 0
    Cohort 2: Interleaving: number analyzed (Participants) | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10
    Cohort 2: Interleaving: Hispanic or Latino |  | 0 |  |  |  |  |  |  |  | 0
    Cohort 2: Interleaving: Not Hispanic or Latino |  | 10 |  |  |  |  |  |  |  | 10
    Cohort 2: Interleaving: Unknown or Not Reported |  | 0 |  |  |  |  |  |  |  | 0
    Cohort 3: Cycling Evolve: number analyzed (Participants) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 4
    Cohort 3: Cycling Evolve: Hispanic or Latino |  |  | 0 |  |  |  |  |  |  | 0
    Cohort 3: Cycling Evolve: Not Hispanic or Latino |  |  | 4 |  |  |  |  |  |  | 4
    Cohort 3: Cycling Evolve: Unknown or Not Reported |  |  | 0 |  |  |  |  |  |  | 0
    Cohort 4: Low Energy Cycling 1: number analyzed (Participants) | 0 | 0 | 0 | 15 | 0 | 0 | 0 | 0 | 0 | 15
    Cohort 4: Low Energy Cycling 1: Hispanic or Latino |  |  |  | 0 |  |  |  |  |  | 0
    Cohort 4: Low Energy Cycling 1: Not Hispanic or Latino |  |  |  | 13 |  |  |  |  |  | 13
    Cohort 4: Low Energy Cycling 1: Unknown or Not Reported |  |  |  | 2 |  |  |  |  |  | 2
    Cohort 5: Low Energy Cycling 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 0 | 0 | 15
    Cohort 5: Low Energy Cycling 2: Hispanic or Latino |  |  |  |  | 0 |  |  |  |  | 0
    Cohort 5: Low Energy Cycling 2: Not Hispanic or Latino |  |  |  |  | 15 |  |  |  |  | 15
    Cohort 5: Low Energy Cycling 2: Unknown or Not Reported |  |  |  |  | 0 |  |  |  |  | 0
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 22 | 0 | 0 | 0 | 22
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Hispanic or Latino |  |  |  |  |  | 1 |  |  |  | 1
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Not Hispanic or Latino |  |  |  |  |  | 21 |  |  |  | 21
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Unknown or Not Reported |  |  |  |  |  | 0 |  |  |  | 0
    Cohort 7: Super Cycle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 0 | 17
    Cohort 7: Super Cycle: Hispanic or Latino |  |  |  |  |  |  | 0 |  |  | 0
    Cohort 7: Super Cycle: Not Hispanic or Latino |  |  |  |  |  |  | 17 |  |  | 17
    Cohort 7: Super Cycle: Unknown or Not Reported |  |  |  |  |  |  | 0 |  |  | 0
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 4
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): Hispanic or Latino |  |  |  |  |  |  |  | 0 |  | 0
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): Not Hispanic or Latino |  |  |  |  |  |  |  | 4 |  | 4
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): Unknown or Not Reported |  |  |  |  |  |  |  | 0 |  | 0
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: Hispanic or Latino |  |  |  |  |  |  |  |  | 0 | 0
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: Not Hispanic or Latino |  |  |  |  |  |  |  |  | 11 | 11
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: Unknown or Not Reported |  |  |  |  |  |  |  |  | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Some participants joined a new cohort once their current cohort was completed, and they met the new cohort guidelines. Therefore, there were participants who ended up in more than one of the 9 cohorts. There were a total of 100 unique participants in this study.
  Participants
    Cohort 1: Low Energy - Continuous: number analyzed (Participants) | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15
    Cohort 1: Low Energy - Continuous: American Indian or Alaska Native | 0 |  |  |  |  |  |  |  |  | 0
    Cohort 1: Low Energy - Continuous: Asian | 0 |  |  |  |  |  |  |  |  | 0
    Cohort 1: Low Energy - Continuous: Black or African American | 1 |  |  |  |  |  |  |  |  | 1
    Cohort 1: Low Energy - Continuous: Native Hawaiian or Other Pacific Islander | 0 |  |  |  |  |  |  |  |  | 0
    Cohort 1: Low Energy - Continuous: White | 14 |  |  |  |  |  |  |  |  | 14
    Cohort 1: Low Energy - Continuous: Other | 0 |  |  |  |  |  |  |  |  | 0
    Cohort 2: Interleaving: number analyzed (Participants) | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10
    Cohort 2: Interleaving: American Indian or Alaska Native |  | 0 |  |  |  |  |  |  |  | 0
    Cohort 2: Interleaving: Asian |  | 0 |  |  |  |  |  |  |  | 0
    Cohort 2: Interleaving: Black or African American |  | 1 |  |  |  |  |  |  |  | 1
    Cohort 2: Interleaving: Native Hawaiian or Other Pacific Islander |  | 0 |  |  |  |  |  |  |  | 0
    Cohort 2: Interleaving: White |  | 9 |  |  |  |  |  |  |  | 9
    Cohort 2: Interleaving: Other |  | 0 |  |  |  |  |  |  |  | 0
    Cohort 3: Cycling Evolve: number analyzed (Participants) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 4
    Cohort 3: Cycling Evolve: American Indian or Alaska Native |  |  | 0 |  |  |  |  |  |  | 0
    Cohort 3: Cycling Evolve: Asian |  |  | 0 |  |  |  |  |  |  | 0
    Cohort 3: Cycling Evolve: Black or African American |  |  | 0 |  |  |  |  |  |  | 0
    Cohort 3: Cycling Evolve: Native Hawaiian or Other Pacific Islander |  |  | 0 |  |  |  |  |  |  | 0
    Cohort 3: Cycling Evolve: White |  |  | 4 |  |  |  |  |  |  | 4
    Cohort 3: Cycling Evolve: Other |  |  | 0 |  |  |  |  |  |  | 0
    Cohort 4: Low Energy Cycling 1: number analyzed (Participants) | 0 | 0 | 0 | 15 | 0 | 0 | 0 | 0 | 0 | 15
    Cohort 4: Low Energy Cycling 1: American Indian or Alaska Native |  |  |  | 1 |  |  |  |  |  | 1
    Cohort 4: Low Energy Cycling 1: Asian |  |  |  | 0 |  |  |  |  |  | 0
    Cohort 4: Low Energy Cycling 1: Black or African American |  |  |  | 3 |  |  |  |  |  | 3
    Cohort 4: Low Energy Cycling 1: Native Hawaiian or Other Pacific Islander |  |  |  | 0 |  |  |  |  |  | 0
    Cohort 4: Low Energy Cycling 1: White |  |  |  | 11 |  |  |  |  |  | 11
    Cohort 4: Low Energy Cycling 1: Other |  |  |  | 0 |  |  |  |  |  | 0
    Cohort 5: Low Energy Cycling 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 0 | 0 | 15
    Cohort 5: Low Energy Cycling 2: American Indian or Alaska Native |  |  |  |  | 0 |  |  |  |  | 0
    Cohort 5: Low Energy Cycling 2: Asian |  |  |  |  | 0 |  |  |  |  | 0
    Cohort 5: Low Energy Cycling 2: Black or African American |  |  |  |  | 1 |  |  |  |  | 1
    Cohort 5: Low Energy Cycling 2: Native Hawaiian or Other Pacific Islander |  |  |  |  | 0 |  |  |  |  | 0
    Cohort 5: Low Energy Cycling 2: White |  |  |  |  | 14 |  |  |  |  | 14
    Cohort 5: Low Energy Cycling 2: Other |  |  |  |  | 0 |  |  |  |  | 0
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 22 | 0 | 0 | 0 | 22
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): American Indian or Alaska Native |  |  |  |  |  | 0 |  |  |  | 0
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Asian |  |  |  |  |  | 0 |  |  |  | 0
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Black or African American |  |  |  |  |  | 0 |  |  |  | 0
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Native Hawaiian or Other Pacific Islander |  |  |  |  |  | 0 |  |  |  | 0
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): White |  |  |  |  |  | 22 |  |  |  | 22
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Other |  |  |  |  |  | 0 |  |  |  | 0
    Cohort 7: Super Cycle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 0 | 17
    Cohort 7: Super Cycle: American Indian or Alaska Native |  |  |  |  |  |  | 0 |  |  | 0
    Cohort 7: Super Cycle: Asian |  |  |  |  |  |  | 0 |  |  | 0
    Cohort 7: Super Cycle: Black or African American |  |  |  |  |  |  | 1 |  |  | 1
    Cohort 7: Super Cycle: Native Hawaiian or Other Pacific Islander |  |  |  |  |  |  | 0 |  |  | 0
    Cohort 7: Super Cycle: White |  |  |  |  |  |  | 16 |  |  | 16
    Cohort 7: Super Cycle: Other |  |  |  |  |  |  | 0 |  |  | 0
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 4
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): American Indian or Alaska Native |  |  |  |  |  |  |  | 0 |  | 0
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): Asian |  |  |  |  |  |  |  | 0 |  | 0
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): Black or African American |  |  |  |  |  |  |  | 0 |  | 0
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): Native Hawaiian or Other Pacific Islander |  |  |  |  |  |  |  | 0 |  | 0
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): White |  |  |  |  |  |  |  | 4 |  | 4
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): Other |  |  |  |  |  |  |  | 0 |  | 0
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: American Indian or Alaska Native |  |  |  |  |  |  |  |  | 0 | 0
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: Asian |  |  |  |  |  |  |  |  | 0 | 0
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: Black or African American |  |  |  |  |  |  |  |  | 1 | 1
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: Native Hawaiian or Other Pacific Islander |  |  |  |  |  |  |  |  | 0 | 0
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: White |  |  |  |  |  |  |  |  | 10 | 10
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: Other |  |  |  |  |  |  |  |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 10 | 4 | 15 | 15 | 22 | 17 | 4 | 11 | 113
Primary Indication [Count of Participants; unit: Participants] — Population: Some participants joined a new cohort once their current cohort was completed, and they met the new cohort guidelines. Therefore, there were participants who ended up in more than one of the 9 cohorts. There were a total of 100 unique participants in this study.
  Participants
    Cohort 1: Low Energy - Continuous: number analyzed (Participants) | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15
    Cohort 1: Low Energy - Continuous: Arachnoiditis | 0 |  |  |  |  |  |  |  |  | 0
    Cohort 1: Low Energy - Continuous: Complex Regional Pain Syndrome | 2 |  |  |  |  |  |  |  |  | 2
    Cohort 1: Low Energy - Continuous: Degenerative Disc Disease | 1 |  |  |  |  |  |  |  |  | 1
    Cohort 1: Low Energy - Continuous: Epidural Fibrosis | 0 |  |  |  |  |  |  |  |  | 0
    Cohort 1: Low Energy - Continuous: Failed Back Surgery Syndrome | 3 |  |  |  |  |  |  |  |  | 3
    Cohort 1: Low Energy - Continuous: Multiple Back Operations | 0 |  |  |  |  |  |  |  |  | 0
    Cohort 1: Low Energy - Continuous: Peripheral Causalgia | 0 |  |  |  |  |  |  |  |  | 0
    Cohort 1: Low Energy - Continuous: Postlaminectomy Pain | 6 |  |  |  |  |  |  |  |  | 6
    Cohort 1: Low Energy - Continuous: Radicular Pain Syndrome | 2 |  |  |  |  |  |  |  |  | 2
    Cohort 1: Low Energy - Continuous: Unsuccessful Disc Surgery | 0 |  |  |  |  |  |  |  |  | 0
    Cohort 1: Low Energy - Continuous: Other | 1 |  |  |  |  |  |  |  |  | 1
    Cohort 2: Interleaving: number analyzed (Participants) | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10
    Cohort 2: Interleaving: Arachnoiditis |  | 0 |  |  |  |  |  |  |  | 0
    Cohort 2: Interleaving: Complex Regional Pain Syndrome |  | 0 |  |  |  |  |  |  |  | 0
    Cohort 2: Interleaving: Degenerative Disc Disease |  | 0 |  |  |  |  |  |  |  | 0
    Cohort 2: Interleaving: Epidural Fibrosis |  | 0 |  |  |  |  |  |  |  | 0
    Cohort 2: Interleaving: Failed Back Surgery Syndrome |  | 0 |  |  |  |  |  |  |  | 0
    Cohort 2: Interleaving: Multiple Back Operations |  | 0 |  |  |  |  |  |  |  | 0
    Cohort 2: Interleaving: Peripheral Causalgia |  | 0 |  |  |  |  |  |  |  | 0
    Cohort 2: Interleaving: Postlaminectomy Pain |  | 5 |  |  |  |  |  |  |  | 5
    Cohort 2: Interleaving: Radicular Pain Syndrome |  | 4 |  |  |  |  |  |  |  | 4
    Cohort 2: Interleaving: Unsuccessful Disc Surgery |  | 0 |  |  |  |  |  |  |  | 0
    Cohort 2: Interleaving: Other |  | 1 |  |  |  |  |  |  |  | 1
    Cohort 3: Cycling Evolve: number analyzed (Participants) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 4
    Cohort 3: Cycling Evolve: Arachnoiditis |  |  | 0 |  |  |  |  |  |  | 0
    Cohort 3: Cycling Evolve: Complex Regional Pain Syndrome |  |  | 0 |  |  |  |  |  |  | 0
    Cohort 3: Cycling Evolve: Degenerative Disc Disease |  |  | 0 |  |  |  |  |  |  | 0
    Cohort 3: Cycling Evolve: Epidural Fibrosis |  |  | 0 |  |  |  |  |  |  | 0
    Cohort 3: Cycling Evolve: Failed Back Surgery Syndrome |  |  | 1 |  |  |  |  |  |  | 1
    Cohort 3: Cycling Evolve: Multiple Back Operations |  |  | 0 |  |  |  |  |  |  | 0
    Cohort 3: Cycling Evolve: Peripheral Causalgia |  |  | 0 |  |  |  |  |  |  | 0
    Cohort 3: Cycling Evolve: Postlaminectomy Pain |  |  | 3 |  |  |  |  |  |  | 3
    Cohort 3: Cycling Evolve: Radicular Pain Syndrome |  |  | 0 |  |  |  |  |  |  | 0
    Cohort 3: Cycling Evolve: Unsuccessful Disc Surgery |  |  | 0 |  |  |  |  |  |  | 0
    Cohort 3: Cycling Evolve: Other |  |  | 0 |  |  |  |  |  |  | 0
    Cohort 4: Low Energy Cycling 1: number analyzed (Participants) | 0 | 0 | 0 | 15 | 0 | 0 | 0 | 0 | 0 | 15
    Cohort 4: Low Energy Cycling 1: Arachnoiditis |  |  |  | 0 |  |  |  |  |  | 0
    Cohort 4: Low Energy Cycling 1: Complex Regional Pain Syndrome |  |  |  | 1 |  |  |  |  |  | 1
    Cohort 4: Low Energy Cycling 1: Degenerative Disc Disease |  |  |  | 3 |  |  |  |  |  | 3
    Cohort 4: Low Energy Cycling 1: Epidural Fibrosis |  |  |  | 0 |  |  |  |  |  | 0
    Cohort 4: Low Energy Cycling 1: Failed Back Surgery Syndrome |  |  |  | 0 |  |  |  |  |  | 0
    Cohort 4: Low Energy Cycling 1: Multiple Back Operations |  |  |  | 0 |  |  |  |  |  | 0
    Cohort 4: Low Energy Cycling 1: Peripheral Causalgia |  |  |  | 0 |  |  |  |  |  | 0
    Cohort 4: Low Energy Cycling 1: Postlaminectomy Pain |  |  |  | 9 |  |  |  |  |  | 9
    Cohort 4: Low Energy Cycling 1: Radicular Pain Syndrome |  |  |  | 1 |  |  |  |  |  | 1
    Cohort 4: Low Energy Cycling 1: Unsuccessful Disc Surgery |  |  |  | 0 |  |  |  |  |  | 0
    Cohort 4: Low Energy Cycling 1: Other |  |  |  | 1 |  |  |  |  |  | 1
    Cohort 5: Low Energy Cycling 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 0 | 0 | 15
    Cohort 5: Low Energy Cycling 2: Arachnoiditis |  |  |  |  | 0 |  |  |  |  | 0
    Cohort 5: Low Energy Cycling 2: Complex Regional Pain Syndrome |  |  |  |  | 0 |  |  |  |  | 0
    Cohort 5: Low Energy Cycling 2: Degenerative Disc Disease |  |  |  |  | 2 |  |  |  |  | 2
    Cohort 5: Low Energy Cycling 2: Epidural Fibrosis |  |  |  |  | 0 |  |  |  |  | 0
    Cohort 5: Low Energy Cycling 2: Failed Back Surgery Syndrome |  |  |  |  | 0 |  |  |  |  | 0
    Cohort 5: Low Energy Cycling 2: Multiple Back Operations |  |  |  |  | 0 |  |  |  |  | 0
    Cohort 5: Low Energy Cycling 2: Peripheral Causalgia |  |  |  |  | 0 |  |  |  |  | 0
    Cohort 5: Low Energy Cycling 2: Postlaminectomy Pain |  |  |  |  | 8 |  |  |  |  | 8
    Cohort 5: Low Energy Cycling 2: Radicular Pain Syndrome |  |  |  |  | 5 |  |  |  |  | 5
    Cohort 5: Low Energy Cycling 2: Unsuccessful Disc Surgery |  |  |  |  | 0 |  |  |  |  | 0
    Cohort 5: Low Energy Cycling 2: Other |  |  |  |  | 0 |  |  |  |  | 0
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 22 | 0 | 0 | 0 | 22
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Arachnoiditis |  |  |  |  |  | 0 |  |  |  | 0
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Complex Regional Pain Syndrome |  |  |  |  |  | 0 |  |  |  | 0
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Degenerative Disc Disease |  |  |  |  |  | 2 |  |  |  | 2
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Epidural Fibrosis |  |  |  |  |  | 0 |  |  |  | 0
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Failed Back Surgery Syndrome |  |  |  |  |  | 2 |  |  |  | 2
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Multiple Back Operations |  |  |  |  |  | 0 |  |  |  | 0
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Peripheral Causalgia |  |  |  |  |  | 0 |  |  |  | 0
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Postlaminectomy Pain |  |  |  |  |  | 14 |  |  |  | 14
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Radicular Pain Syndrome |  |  |  |  |  | 4 |  |  |  | 4
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Unsuccessful Disc Surgery |  |  |  |  |  | 0 |  |  |  | 0
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Other |  |  |  |  |  | 0 |  |  |  | 0
    Cohort 7: Super Cycle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 0 | 17
    Cohort 7: Super Cycle: Arachnoiditis |  |  |  |  |  |  | 0 |  |  | 0
    Cohort 7: Super Cycle: Complex Regional Pain Syndrome |  |  |  |  |  |  | 0 |  |  | 0
    Cohort 7: Super Cycle: Degenerative Disc Disease |  |  |  |  |  |  | 1 |  |  | 1
    Cohort 7: Super Cycle: Epidural Fibrosis |  |  |  |  |  |  | 0 |  |  | 0
    Cohort 7: Super Cycle: Failed Back Surgery Syndrome |  |  |  |  |  |  | 2 |  |  | 2
    Cohort 7: Super Cycle: Multiple Back Operations |  |  |  |  |  |  | 0 |  |  | 0
    Cohort 7: Super Cycle: Peripheral Causalgia |  |  |  |  |  |  | 0 |  |  | 0
    Cohort 7: Super Cycle: Postlaminectomy Pain |  |  |  |  |  |  | 9 |  |  | 9
    Cohort 7: Super Cycle: Radicular Pain Syndrome |  |  |  |  |  |  | 3 |  |  | 3
    Cohort 7: Super Cycle: Unsuccessful Disc Surgery |  |  |  |  |  |  | 0 |  |  | 0
    Cohort 7: Super Cycle: Other |  |  |  |  |  |  | 2 |  |  | 2
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 4
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): Arachnoiditis |  |  |  |  |  |  |  | 0 |  | 0
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): Complex Regional Pain Syndrome |  |  |  |  |  |  |  | 0 |  | 0
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): Degenerative Disc Disease |  |  |  |  |  |  |  | 1 |  | 1
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): Epidural Fibrosis |  |  |  |  |  |  |  | 0 |  | 0
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): Failed Back Surgery Syndrome |  |  |  |  |  |  |  | 1 |  | 1
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): Multiple Back Operations |  |  |  |  |  |  |  | 0 |  | 0
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): Peripheral Causalgia |  |  |  |  |  |  |  | 0 |  | 0
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): Postlaminectomy Pain |  |  |  |  |  |  |  | 0 |  | 0
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): Radicular Pain Syndrome |  |  |  |  |  |  |  | 2 |  | 2
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): Unsuccessful Disc Surgery |  |  |  |  |  |  |  | 0 |  | 0
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): Other |  |  |  |  |  |  |  | 0 |  | 0
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: Arachnoiditis |  |  |  |  |  |  |  |  | 0 | 0
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: Complex Regional Pain Syndrome |  |  |  |  |  |  |  |  | 2 | 2
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: Degenerative Disc Disease |  |  |  |  |  |  |  |  | 0 | 0
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: Epidural Fibrosis |  |  |  |  |  |  |  |  | 0 | 0
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: Failed Back Surgery Syndrome |  |  |  |  |  |  |  |  | 0 | 0
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: Multiple Back Operations |  |  |  |  |  |  |  |  | 0 | 0
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: Peripheral Causalgia |  |  |  |  |  |  |  |  | 0 | 0
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: Postlaminectomy Pain |  |  |  |  |  |  |  |  | 8 | 8
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: Radicular Pain Syndrome |  |  |  |  |  |  |  |  | 1 | 1
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: Unsuccessful Disc Surgery |  |  |  |  |  |  |  |  | 0 | 0
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: Other |  |  |  |  |  |  |  |  | 0 | 0
Years Since Onset of Chronic Pain [Mean (Standard Deviation); unit: years] — Population: Some participants joined a new cohort once their current cohort was completed, and they met the new cohort guidelines. Therefore, there were participants who ended up in more than one of the 9 cohorts. There were a total of 100 unique participants in this study.
  years
    Cohort 1: Low Energy - Continuous: number analyzed (Participants) | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15
    Cohort 1: Low Energy - Continuous | 13.7 (9.8) |  |  |  |  |  |  |  |  | 13.7 (9.8)
    Cohort 2: Interleaving: number analyzed (Participants) | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10
    Cohort 2: Interleaving |  | 21.5 (15.8) |  |  |  |  |  |  |  | 21.5 (15.8)
    Cohort 3: Cycling Evolve: number analyzed (Participants) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 4
    Cohort 3: Cycling Evolve |  |  | 27.0 (18.7) |  |  |  |  |  |  | 27.0 (18.7)
    Cohort 4: Low Energy Cycling 1: number analyzed (Participants) | 0 | 0 | 0 | 15 | 0 | 0 | 0 | 0 | 0 | 15
    Cohort 4: Low Energy Cycling 1 |  |  |  | 20.7 (16.4) |  |  |  |  |  | 20.7 (16.4)
    Cohort 5: Low Energy Cycling 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 0 | 0 | 15
    Cohort 5: Low Energy Cycling 2 |  |  |  |  | 16.5 (8.4) |  |  |  |  | 16.5 (8.4)
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 22 | 0 | 0 | 0 | 22
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS) |  |  |  |  |  | 20.6 (12.4) |  |  |  | 20.6 (12.4)
    Cohort 7: Super Cycle: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 0 | 17
    Cohort 7: Super Cycle |  |  |  |  |  |  | 9.5 (9.1) |  |  | 9.5 (9.1)
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 4
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS) |  |  |  |  |  |  |  | 4.25 (2.6) |  | 4.25 (2.6)
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow |  |  |  |  |  |  |  |  | 17.8 (17.17) | 17.8 (17.17)
Days Since Implant to Enrollment [Mean (Standard Deviation); unit: days] — Population: Some participants joined a new cohort once their current cohort was completed, and they met the new cohort guidelines. Therefore, there were participants who ended up in more than one of the 9 cohorts. There were a total of 100 unique participants in this study.
  days
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 0 | 17
    (all) |  |  |  |  |  |  | 13.9 (3.8) |  |  | 13.9 (3.8)
Years Since Implant to Enrollment [Mean (Standard Deviation); unit: years] — Population: Some participants joined a new cohort once their current cohort was completed, and they met the new cohort guidelines. Therefore, there were participants who ended up in more than one of the 9 cohorts. There were a total of 100 unique participants in this study.
  years
    Cohort 1: Low Energy - Continuous: number analyzed (Participants) | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15
    Cohort 1: Low Energy - Continuous | 0.9 (1.0) |  |  |  |  |  |  |  |  | 0.9 (1.0)
    Cohort 2: Interleaving: number analyzed (Participants) | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10
    Cohort 2: Interleaving |  | 0.8 (0.4) |  |  |  |  |  |  |  | 0.8 (0.4)
    Cohort 3: Cycling Evolve: number analyzed (Participants) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 4
    Cohort 3: Cycling Evolve |  |  | 1.1 (0.5) |  |  |  |  |  |  | 1.1 (0.5)
    Cohort 4: Low Energy Cycling 1: number analyzed (Participants) | 0 | 0 | 0 | 15 | 0 | 0 | 0 | 0 | 0 | 15
    Cohort 4: Low Energy Cycling 1 |  |  |  | 1.1 (0.5) |  |  |  |  |  | 1.1 (0.5)
    Cohort 5: Low Energy Cycling 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 0 | 0 | 15
    Cohort 5: Low Energy Cycling 2 |  |  |  |  | 1.1 (0.5) |  |  |  |  | 1.1 (0.5)
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 22 | 0 | 0 | 0 | 22
    Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS) |  |  |  |  |  | 1.6 (1.0) |  |  |  | 1.6 (1.0)
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 4
    Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS) |  |  |  |  |  |  |  | 0.83 (0.4) |  | 0.83 (0.4)
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11
    Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow |  |  |  |  |  |  |  |  | 4.5 (4.37) | 4.5 (4.37)

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Rating Scale (NPRS) - Cohort 1
Description: To characterize the effect of different programmed settings on pain relief. The NPRS will be recorded once or daily over a period of time, where the subjects will rate their pain on a 11-point numeric rating scale of 0 to 10, with 0 representing 'No Pain' and 10 representing 'Worst pain imaginable'. The average overall NPRS pain score prior to the scheduled visit will be used for analysis.
Time Frame: Up to 5 months
Population: Number analyzed refers to patients with measure available.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cohort 1: Low Energy - Continuous Initial: Subjects will be programmed to a specific frequency with a long pulse width at various amplitudes
  Spinal Cord Stimulation: Programming
Arm/Group | Cohort 1: Low Energy - Continuous Initial
Number analyzed (Participants) | 14
score on a scale
  Enrollment | 5.2 (2.5)
  Comfortable amplitude (Period 1): number analyzed (Participants) | 13
  Comfortable amplitude (Period 1) | 4.9 (2.3)
  80% comfortable amplitude (Period 2): number analyzed (Participants) | 13
  80% comfortable amplitude (Period 2) | 5.1 (2.3)
  60% comfortable amplitude (Period 3): number analyzed (Participants) | 12
  60% comfortable amplitude (Period 3) | 4.9 (2.1)
  40% comfortable amplitude (Period 4): number analyzed (Participants) | 12
  40% comfortable amplitude (Period 4) | 4.6 (2.1)
  20% comfortable amplitude (Period 5): number analyzed (Participants) | 11
  20% comfortable amplitude (Period 5) | 4.7 (2.0)
  0 mA/V (Period 6): number analyzed (Participants) | 11
  0 mA/V (Period 6) | 4.7 (1.9)
  Comfortable amplitude with 25% duty cycle (Period 7): number analyzed (Participants) | 11
  Comfortable amplitude with 25% duty cycle (Period 7) | 4.3 (2.3)
  The "best" amplitude and cycling enabling 5 years on a PC (Period 8): number analyzed (Participants) | 10
  The "best" amplitude and cycling enabling 5 years on a PC (Period 8) | 4.7 (1.9)

2. Primary Outcome: Numeric Pain Rating Scale (NPRS) - Cohort 2
Description: as for outcome 1
Time Frame: Up to 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 2: Interleaving
Number analyzed (Participants) | 9
score on a scale
  Enrollment | 4.6 (2.46)
  Follow-up (HD) | 4.3 (2.48)
  Follow-up (LD) | 5.5 (1.33)

3. Primary Outcome: Numeric Pain Rating Scale (NPRS) - Cohort 3
Description: as for outcome 1
Time Frame: Up to 3 months
Population: Number analyzed refers to patients with measure available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 3: Cycling Evolve
Number analyzed (Participants) | 4
score on a scale
  Enrollment | 4.0 (2.6)
  Follow Up 1 (Came in at Cycling Off) | 3.9 (2.4)
  Follow Up 2 (Came in at Cycling ON) | 4.9 (2.2)
  Follow Up 3 (Came in at Cycling ON) | 4.5 (2.1)
  Follow Up 4 (Came in at Cycling ON) | 4.7 (2.5)
  Follow Up 5 (Came in at Cycling ON) | 4.2 (2.4)
  Final Study Visit (Came in at Cycling ON): number analyzed (Participants) | 3
  Final Study Visit (Came in at Cycling ON) | 3.2 (2.2)

4. Primary Outcome: Numeric Pain Rating Scale (NPRS) - Cohort 4
Description: as for outcome 1
Time Frame: Up to 5 months
Population: Number analyzed refers to patients with measure available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 4: Low Energy Cycling 1
Number analyzed (Participants) | 15
score on a scale
  Enrollment | 3.9 (3.0)
  Low Energy 1, cycling off (Period 1) | 4.9 (2.4)
  Low Energy 1, cycling ON (Period 2) | 5.1 (2.0)
  Low Energy 1, cycling ON (Period 3): number analyzed (Participants) | 14
  Low Energy 1, cycling ON (Period 3) | 5.6 (2.1)
  Low Energy 2, cycling off (Period 4): number analyzed (Participants) | 14
  Low Energy 2, cycling off (Period 4) | 4.7 (2.3)
  Low Energy 2, cycling ON (Period 5): number analyzed (Participants) | 13
  Low Energy 2, cycling ON (Period 5) | 4.9 (2.3)
  Low Energy 2, cycling ON (Period 6): number analyzed (Participants) | 13
  Low Energy 2, cycling ON (Period 6) | 5.1 (2.4)
  Low Energy 2, cycling ON (Period 7): number analyzed (Participants) | 13
  Low Energy 2, cycling ON (Period 7) | 5.3 (2.4)

5. Primary Outcome: Numeric Pain Rating Scale - Cohort 5
Description: as for outcome 1
Time Frame: Up to 5 months
Population: Number analyzed refers to patients with measure available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 5: Low Energy Cycling 2
Number analyzed (Participants) | 15
score on a scale
  Enrollment | 4.8 (2.5)
  Low Energy 1, cycling off (Period 1) | 5.0 (1.9)
  Low Energy 1, cycling ON (Period 2) | 5.0 (2.0)
  Low Energy 1, cycling ON (Period 3) | 5.2 (2.3)
  Low Energy 2, cycling off (Period 4): number analyzed (Participants) | 14
  Low Energy 2, cycling off (Period 4) | 4.2 (2.0)
  Low Energy 2, cycling ON (Period 5): number analyzed (Participants) | 14
  Low Energy 2, cycling ON (Period 5) | 4.7 (2.2)
  Low Energy 2, cycling ON (Period 6): number analyzed (Participants) | 13
  Low Energy 2, cycling ON (Period 6) | 4.5 (1.8)

6. Primary Outcome: Numeric Pain Rating Scale (NPRS) - Cohort 6
Description: as for outcome 1
Time Frame: Up to 7 months
Population: Number analyzed refers to patients with measure available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS)
Number analyzed (Participants) | 22
score on a scale
  Enrollment | 3.5 (1.8)
  Washout (Follow-up 1): number analyzed (Participants) | 21
  Washout (Follow-up 1) | 5.6 (2.0)
  DTM-LE Continuous (Follow-up 2) | 4.3 (2.1)
  DTM-LE Duty Cycle Enabled* (Follow-up 3): number analyzed (Participants) | 21
  DTM-LE Duty Cycle Enabled* (Follow-up 3) | 4.4 (2.1)
  2-Week Follow-up (Follow-up 4): number analyzed (Participants) | 20
  2-Week Follow-up (Follow-up 4) | 3.7 (1.6)
  1-Month Follow-up (Follow-up 5): number analyzed (Participants) | 19
  1-Month Follow-up (Follow-up 5) | 3.8 (1.7)
  2-Month Follow-up (Follow-up 6): number analyzed (Participants) | 20
  2-Month Follow-up (Follow-up 6) | 4.2 (1.1)
  3-Month Follow-up (Final Study Visit): number analyzed (Participants) | 20
  3-Month Follow-up (Final Study Visit) | 4.0 (1.4)

7. Primary Outcome: Numeric Pain Rating Scale (NPRS) - Cohort 7
Description: as for outcome 1
Time Frame: Up to 8 months
Population: Number analyzed refers to patients with measure available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 7: Super Cycle
Number analyzed (Participants) | 17
score on a scale
  Pre-SCS Pain Score | 8.5 (1.4)
  Enrollment | 5.5 (3.0)
  Optimization Visit 1 (Follow Up 1): number analyzed (Participants) | 15
  Optimization Visit 1 (Follow Up 1) | 6.1 (2.2)
  Optimization Visit 2 (Follow Up 2): number analyzed (Participants) | 14
  Optimization Visit 2 (Follow Up 2) | 5.2 (2.2)
  Optimization Visit 3 (Follow Up 3): number analyzed (Participants) | 12
  Optimization Visit 3 (Follow Up 3) | 4.2 (2.0)
  Start of Titration Phase (Follow Up 4): number analyzed (Participants) | 11
  Start of Titration Phase (Follow Up 4) | 4.0 (2.0)
  2-Week Titration Phase (Follow Up 5): number analyzed (Participants) | 8
  2-Week Titration Phase (Follow Up 5) | 4.6 (2.3)
  4-Week Titration Phase (Follow Up 6): number analyzed (Participants) | 7
  4-Week Titration Phase (Follow Up 6) | 3.6 (2.3)
  End of Titration Phase (Follow Up 7): number analyzed (Participants) | 6
  End of Titration Phase (Follow Up 7) | 3.2 (1.7)
  1-Month Post Titration Phase (Follow Up 8): number analyzed (Participants) | 6
  1-Month Post Titration Phase (Follow Up 8) | 3.3 (2.1)
  2-Months Post Titration Phase (Follow Up 9): number analyzed (Participants) | 6
  2-Months Post Titration Phase (Follow Up 9) | 4.3 (3.1)
  3-Months Post Titration Phase (Final Study Visit): number analyzed (Participants) | 6
  3-Months Post Titration Phase (Final Study Visit) | 3.0 (3.1)

8. Primary Outcome: Numeric Pain Rating Scale (NPRS) - Cohort 8
Description: as for outcome 1
Time Frame: Up to 0.5 months
Population: Number analyzed refers to patients with measure available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS)
Number analyzed (Participants) | 4
score on a scale
  Enrollment | 3 (1.83)
  Final Study Visit | 3.25 (2.22)

9. Primary Outcome: Numeric Pain Rating Scale at Enrollment (NPRS) - Cohort 9
Description: as for outcome 1
Time Frame: Up to 1 month
Population: Number analyzed refers to patients with measure available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow
Number analyzed (Participants) | 10
score on a scale | 3.8 (2.25)

ADVERSE EVENTS:
Time Frame: Cohort 1: 4.4 months Cohort 2: 1.5 months Cohort 3: 3.0 months Cohort 4: 2.1 months Cohort 5: 2.8 months Cohort 6: 6.8 months Cohort 7: 7.8 months Cohort 8: 0.5 months Cohort 9: 0.6 months
Groups:
- Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS): Effects of decreased frequency and therapy cycling parameters Spinal Cord Stimulation: Programming
Arm/Group | Cohort 1: Low Energy - Continuous | Cohort 2: Interleaving | Cohort 3: Cycling Evolve | Cohort 4: Low Energy Cycling 1 | Cohort 5: Low Energy Cycling 2 | Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS) | Cohort 7: Super Cycle | Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS) | Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/10 | 0/4 | 0/15 | 0/15 | 0/22 | 0/17 | 0/4 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/10 | 0/4 | 0/15 | 0/15 | 0/22 | 0/17 | 0/4 | 0/11
Other Adverse Events (participants affected / at risk) | 5/15 | 1/10 | 0/4 | 4/15 | 2/15 | 3/22 | 3/17 | 0/4 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Low Energy - Continuous (N=15) | Cohort 2: Interleaving (N=10) | Cohort 3: Cycling Evolve (N=4) | Cohort 4: Low Energy Cycling 1 (N=15) | Cohort 5: Low Energy Cycling 2 (N=15) | Cohort 6: Differential Targeted Multiplexed-Low Energy Spinal Cord Stimulation (DTM-LE SCS) (N=22) | Cohort 7: Super Cycle (N=17) | Cohort 8: Differential Targeted Multiplexed (DTM) for Neuro Sense (NS) (N=4) | Cohort 9: Diabetic Peripheral Neuropathy (DPN) Flow (N=11)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Pain (General disorders) | 3 (3) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | NA | 1 (1) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Device stimulation issue (Product Issues) | 0 (0) | 0 (0) | NA | 3 (4) | 2 (2) | 0 (0) | 0 (0) | NA | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Headache (Nervous system disorders) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Medical device site irritation (General disorders) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Medical device site pain (General disorders) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT03763708/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT03763708/SAP_001.pdf